CLINICAL TRIAL: NCT04449068
Title: Pre et Post-operative Evaluation of Patients With Tourette Syndrome Treated With High Frequency Bilateral Stimulation of the Anterior Part of the Internal Pallid Globus
Brief Title: Observational Database on Deep Brain Stimulation in Tourette Syndrome
Acronym: POSTSTIC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190808
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Tourette Syndrome
Keywords: bilateral deep brain stimulation; Tourette syndrome,
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of patients with Tourette's Gilles Syndrome: Neurological and neuropsychological evaluations of patients with Tourette's Gilles syndrome treated with high frequency bilateral stimulation of the anterior part of the internal pallid globus
  Interventions: Other: Neurological and neuropsychological Follow-up after deep brain stimulation

INTERVENTIONS:
Other: Neurological and neuropsychological Follow-up after deep brain stimulation — Investigation of tic severity, psychiatric co-morbidities, quality of life, and neuropsychologcial measures until the 5-year after deep brain stimulation (DBS)

SUMMARY:
Within an ongoing deep brain stimulation (DBS) program for Tourette syndrome (TS) at the Department of Neurology, Pitié-Salpêtrière Hospital, Paris/France, the investigator team plans to evaluate patients pre-operatively and then at one year intervals post-operatively until the 5-year mark has been achieved. The investigator team will investigate tic severity, psychiatric co-morbidities, quality of life, and neuropsychological measures.

DETAILED DESCRIPTION:
Since the completion of the STIC trial in 2017, the french team continues to offer DBS of the globus pallidus internus (GPi) to selected, treatment-refractory patients with TS. On average, three to four patients undergo surgery every year. Even though a first follow-up of the STIC cohort up to four years post-op indicates ongoing improvement of tic severity, many questions remains regarding the efficacy of GPi DBS in TS. These questions include frequent comorbidities of TS, quality of life, evolution of medication and stimulation parameters, as well as neuropsychological functioning. Therefore, the investigator proposes to evaluate all patients undergoing GPi DBS for TS to be evaluated comprehensively pre-operatively and once yearly after surgery until reaching the 5-year mark. The investigator team hopes these data may help to plan for future international multicenter trials, and provide indications on prognostic factors concerning response to GPi DBS in TS.

ELIGIBILITY:
Inclusion Criteria:

* Tourette syndrome severe and drug-resistant eligible for bilateral deep brain stimulation
* Person who voluntarily and knowledgeably agreed to participate in the study

Exclusion Criteria:

* Non affiliation to a French social security system (recipient or assign) excluding AME

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Tourette syndrome eligible for bilateral deep brain stimulation of the anterior internal pallid globus
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2031-06-12 (Estimated); Study Completion 2031-06-12 (Estimated)

PRIMARY OUTCOMES:
Measure the severity of tics | Month 60
  Measure the severity of tics, determined by the YGTSS-R (Yale Global Tic Severity Scale score - revised) .
  The overall score is between 0 (no TICS) and 100 (severity in TICS) therefore a score decrease is expected .

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Neurosciences, GH Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Welter ML, Houeto JL, Thobois S, Bataille B, Guenot M, Worbe Y, Hartmann A, Czernecki V, Bardinet E, Yelnik J, du Montcel ST, Agid Y, Vidailhet M, Cornu P, Tanguy A, Ansquer S, Jaafari N, Poulet E, Serra G, Burbaud P, Cuny E, Aouizerate B, Pollak P, Chabardes S, Polosan M, Borg M, Fontaine D, Giordana B, Raoul S, Rouaud T, Sauvaget A, Jalenques I, Karachi C, Mallet L; STIC study group. Anterior pallidal deep brain stimulation for Tourette's syndrome: a randomised, double-blind, controlled trial. Lancet Neurol. 2017 Aug;16(8):610-619. doi: 10.1016/S1474-4422(17)30160-6. Epub 2017 Jun 20. PMID 28645853
- [Background] Welter ML, Houeto JL, Worbe Y, Diallo MH, Hartmann A, Tezenas du Montcel S, Ansquer S, Thobois S, Fontaine D, Rouaud T, Cuny E, Karachi C, Mallet L; STIC study group. Long-term effects of anterior pallidal deep brain stimulation for tourette's syndrome. Mov Disord. 2019 Apr;34(4):586-588. doi: 10.1002/mds.27645. Epub 2019 Feb 20. No abstract available. PMID 30788865